CLINICAL TRIAL: NCT01637584
Title: Neurobiology of Sleep and Sleep Treatment Response in Returning Veterans
Acronym: NOSSTIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Anne Germain, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO08050307
Record Dates: First submitted 2012-06-15; First posted 2012-07-11 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-03

CONDITIONS: Non PTSD; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prazosin (Experimental): Active medication arm. Prazosin is an FDA approved medication, originally designed as an anti-hypertension medication. Side effects of the medication in some include sleepiness and once asleep, sustained sleep.
  Interventions: Drug: Prazosin
- Placebo (Placebo Comparator): A placebo is a sugar pill, which will be used to compare with the results of the active medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prazosin — The medication will be administered in the same manner, regardless of active or placebo, as the study physician and investigators, as well as the participants, will be blind to the type of medication they are taking.
  Arms: Prazosin
Drug: Placebo — The medication will be administered in the same manner, regardless of active or placebo, as the study physician and investigators, as well as the participants, will be blind to the type of medication they are taking.
  Arms: Placebo

SUMMARY:
The overarching objectives of this study are: 1) To investigate the neurobiology of posttraumatic stress disorder (PTSD) during Rapid Eye Movement (REM) and Non-Rapid Eye Movement (NREM) sleep relative to wakefulness; 2) To identify the neurobiological underpinnings of sleep treatment response to prazosin or placebo during wakefulness, REM sleep, and NREM sleep in Operation Iraqi Freedom/Operation Enduring Freedom (OIF/OEF) ( veterans with PTSD; and 3) To explore pre-treatment brain activity patterns during wakefulness, REM sleep, and NREM sleep that predict sleep treatment response. We will also explore the stability of the Positron Emission Tomography (PET) signal by comparing pre- and post-placebo changes in brain glucose metabolism in non-responders. For non-PTSD veterans, the stability of the PET signal will be evaluated in a subsample of 6 veterans without PTSD who will repeat the PET imaging procedures 8 weeks after the initial PET series.

The overarching hypothesis is that PTSD is characterized by neurobiological alterations in the amygdala, medial prefrontal cortex (mPFC), and brain centers involved in the regulation of NREM and REM sleep, and that these neurobiological changes are normalized with effective sleep treatment.

DETAILED DESCRIPTION:
PTSD affects both daytime functioning and sleep. Complaints of poor sleep, objective disruption of sleep, and heightened sympathovagal tone during sleep occurring early after trauma exposure increase the risk of developing PTSD up to one year later. (1-4). Insomnia is one the most common reasons for referral to mental health services in active duty personnel (5). In military personnel returning from Iraq and Afghanistan, more than 70 percent of those with PTSD report sleep problems and fatigue, whereas more than 25% percent of those without PTSD endorse these symptoms (6). Other disruptive nocturnal behaviors and sleep disorders including sleep terrors, nocturnal anxiety attacks, simple and complex motor behaviors and vocalizations, acting out dreams, sleep apnea, and periodic leg movement disorders are also frequently reported by PTSD patients (7-12). In PTSD, sleep disturbances independently contribute to poor clinical outcomes such as increased severity of daytime PTSD symptoms (8), depression (13), suicidality (13), general psychiatric distress (14), poorer quality of life and functioning (14), poorer perceived physical health (14), and increased substance use (15;16).

ELIGIBILITY:
Inclusion Criteria:

* OIF/OEF veteran
* Between the ages of 18 and 50 years old
* Not taking medications known to affect sleep or wake function for 2 weeks

Additional selection criteria for PTSD subjects are:

* Trauma occurred three months or more before study entry
* Meeting diagnostic criteria for current PTSD according to the Clinician Administered PTSD Scale (CAPS)
* Participants will remain in ongoing counseling services

Additional selection criterion for non-PTSD healthy subjects:

* Not meet DSM-IV diagnostic criteria for current PTSD
* Have a total score < 13 on the Beck Depression Inventory
* Participants who are active-duty military personnel will be required to obtain permission from their commander to participate in this study.

Exclusion Criteria:

* Current diagnosis of untreated, severe depression as determined by the Structured Clinical Interview for Diagnostic and Statistical Manual- IV Edition (DSM-IV), non-patient version
* Beck Depression Inventory > 30
* History of psychotic or bipolar disorder
* Current history (within 3 months) of substance or alcohol abuse
* Significant or unstable acute or chronic medical conditions
* Other current sleep disorders
* Presence of implanted devices or metal in body such as cardiac pacemaker, aneurysm clip, ear implant, shrapnel, neurostimulators or other metal devices
* Fear of closed spaces
* Previous radiation exposure (past year) that exceeds recommended safety limits
* Pregnancy or breast feeding
* Resting blood pressure < 90/60 at the screening physical examination
* Heart rate > 100 beats/minutes
* Current use of a beta-blocker
* Use of an alpha-1 antagonist agent in the previous 3 weeks
* Refusal to follow the safety measures in the case of use of a phosphodiesterase 5 inhibitor (Cialis, Viagra, Levitra)
* Unexpected, untreated, or serious EKG findings

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Stocker RP, Cieply MA, Paul B, Khan H, Henry L, Kontos AP, Germain A. Combat-related blast exposure and traumatic brain injury influence brain glucose metabolism during REM sleep in military veterans. Neuroimage. 2014 Oct 1;99:207-14. doi: 10.1016/j.neuroimage.2014.05.067. Epub 2014 Jun 2. PMID 24893322

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prazosin | Placebo
Started | 20 | 20
Completed | 19 | 17
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: Comparison on demographic variables
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (6.55) | 27.2 (6.25) | 27.7 (5.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Whole Brain Relative Regional Cerebral Metabolic Rate of Glucose
Description: The reported Z value reflect the magnitude of the state difference (Wake vs. Non-REM or Wake vs. REM) within the prazosin group pre-to-post treatment, and after using a mask to adjust for the spurious effects of the passage of time.
Time Frame: Baseline and post-intervention at 8-10 weeks
Population: 9 of the 20 participants who were randomized to prazosin and 13 of the participants randomized to placebo provided scans pre- and post-treatment that were of sufficiency quality to be included in the final analyses.
Measure: Number; unit: Z values
Groups:
- Prazosin -Placebo: Difference in relative brain glucose metabolism between states and pre-to-post treatment for participants randomized to prazosin after adjusting for non-significant changes in the placebo group.
Arm/Group | Prazosin -Placebo
Number analyzed (Participants) | 22
Z values
  Pre-to-Post Treatment (Wakefulness > NREM) | 3.78
  Pre-to-Post Treatment (Wakefulness < NREM) | 3.76
  Pre-to-Post Treatment (Wakefulness > REM) | 3.52
  Pre-to-Post Treatment (Wakefulness < REM) | 3.36
  Within-state time-dependent decrease in rCMRglc | 4.12
  Within-state time-dependent increase in rCMRglc | 3.89
Statistical Analysis 1: Comparison: Prazosin -Placebo; Wakefulness > Non-Rapid Eye Movement (NREM): Mean K-cluster voxels (Ke)=15,586: x,y,z= -36, -74, 0. Left Brodmann's Area (BA) 3, 6, 7, 10, 17, 19, 20,21,23, 38; Test type: Superiority or Other; p < 0.001, Full Factorial ANOVAs and Paired T-tests — Threshold for significance: <.05
Statistical Analysis 2: Comparison: Prazosin -Placebo; Wakefulness < NREM: Ke=7,013: x,y,z= 26, 22, -40. Right BA 4, 10-14, 21, 25, 32, 38, 45;; Test type: Superiority or Other; p = 0.039, Full Factorial ANOVAs and Paired T-tests — Threshold for significance: <.05
Statistical Analysis 3: Comparison: Prazosin -Placebo; Wakefulness > (Rapid Eye Movement (REM): No cluster size, coordinates, or brain regions to report; Test type: Superiority or Other; p = 0.701, Full Factorial ANOVAs and Paired T-tests — Threshold for significance: <.05
Statistical Analysis 4: Comparison: Prazosin -Placebo; Wakefulness < REM: No cluster size, coordinates, or brain regions to report; Test type: Superiority or Other; p = 1.00, Full Factorial ANOVAs and Paired T-tests — Threshold for significance: <.05
Statistical Analysis 5: Comparison: Prazosin -Placebo; Within-state decrease in rCMRglc: Ke=6,150: x,y,z= -30, -30, 2. Left BA 40, insula, hippocampus, caudate, and putamen;; Test type: Superiority or Other; p = 0.03, Full Factorial ANOVAs and Paired T-tests — Threshold for significance: <.05
Statistical Analysis 6: Comparison: Prazosin -Placebo; Within-state increase in rCMRglc: Ke=7,049: x,y,z= 66, -18, 26. Right BA 1, 3, 15, 21, 22, 23, 41, 42; Test type: Superiority or Other; p = 0.01, Full Factorial ANOVAs and Paired T-tests — Threshold for significance: <.05

2. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI):
Description: Self-report sleep quality measure. Scores range from 0 to 21, with higher scores reflecting poorer sleep quality.
Time Frame: Baseline and post-treatment at 8-10 weeks
Population: 9 of the 20 participants who were randomized to prazosin and 13 of the participants randomized to prazosin provided scans pre- and post-treatment that were of sufficiency quality to be included in the final analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 9 | 13
units on a scale
  PSQI: Baseline | 9.25 (2.64) | 8.08 (2.72)
  PSQI: Post | 6.71 (4.31) | 6.54 (2.57)

ADVERSE EVENTS:
Arm/Group | Prazosin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No